CLINICAL TRIAL: NCT02947295
Title: Global Genomic and Proteomic Profiling of African Children With Typhoid Fever
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0445-12 EP
Record Dates: First submitted 2014-12-01; First posted 2016-10-27 (Estimated); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Typhoid Fever
MeSH Terms: conditions — Typhoid Fever

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, stool, nasopharyngeal swab/aspirate as well as cerebrospinal fluid (CSF), pleural fluid, induced sputum, gastric aspirates or synovial fluid with clinical indication.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To develop a rapid, sensitive, and inexpensive diagnostic method, as well as more efficacious vaccine, for countries where typhoid fever remains a major public health burden.

DETAILED DESCRIPTION:
Typhoid fever is caused by Salmonella enteric serovar Typhi (S. typhi), a human specific pathogen. The World Health Organization (WHO) recognizes typhoid fever as a global health problem, with an estimated 21 million cases and 200,000-600,000 deaths annually. In Africa and South Asia, young children represent a subgroup with the highest disease burden. The onset of the illness is insidious and clinical diagnosis is often unreliable. Definitive diagnosis through blood or bone-marrow culture is labor-intensive, expensive, and invasive, with a sensitivity of 40 to 70%. WHO recommends routine typhoid fever vaccination but currently licensed vaccines provide only 55-75% protection against the disease. Therefore, there is an urgent need to develop rapid, sensitive, and inexpensive diagnostic methods, as well as more efficacious vaccines for countries where typhoid fever remains a major public health burden. The long term goals are 1) to develop innovative molecular diagnostic assays for rapid and inexpensive detection of typhoid fever and, 2) to better understand the molecular mechanisms of host response to facilitate the development of next-generation typhoid fever vaccines.

The immediate objective is to obtain global gene expression and proteomic profiles of S. Typhi infected African children, identify and validate the classifier genes and proteins as potential diagnostic biomarkers and vaccine targets. A bacteremia surveillance system was established in central Nigeria in 2008; a pilot study was initiated from a small cohort from this system composed of children with typhoid fever.

Preliminary data showed unique gene expression profiles of host response in peripheral blood of children with typhoid fever compared with other bacteremic infections, as well as patients in acute vs. convalescent phase. Here, it is hypothesized that distinct classifier genes and proteins based on host response in the peripheral blood and serum can be obtained to discriminate typhoid fever from other bacteremic infections and healthy controls.

Specific aims:

1. Define typhoid fever-specific host response classifier genes using gene expression (GE) micro-arrays,
2. Discover specific serum anti-typhoid fever proteins using newly established S. Typhi proteome micro-arrays and develop prototype serologic assay for acute typhoid (ELISA)
3. Validate classifier genes and field-test prototype ELISAs using new, independent cohorts.

To accomplish these objectives, a multidisciplinary team with expertise in infectious disease, immunology, molecular genomics/proteomics, micro-arrays, and bioinformatics has been assembled to ensure success of this project. These studies will identify distinct classifier genes and proteins of typhoid fever infection based on immunological responses. Classifiers that discriminate S. Typhi from other bacteremia are possible to develop and offer rapid, inexpensive, non-invasive, and sensitive molecular diagnostic assays specific for typhoid fever. Classifier proteins obtained from the new, custom whole-proteome typhoid fever micro-arrays will provide new insights of targeted proteins and antibodies for next-generation vaccine development.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 1-14 years who present with an acute febrile illness that is clinically suggestive of bacteremia.

Exclusion Criteria:

* Children who have underlying conditions that are recognized to increase susceptibility to invasive salmonellosis. Other conditions that are associated with frequent opportunistic infections that may cause aberrations of immune function will also be excluded, such as human immunodeficiency virus (HIV) infection and malnutrition. Clinical conditions that are known to be associated with increased risk of salmonella carriage will also be excluded, such as schistosomiasis.

Ages: 1 Minute to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children 1-14 years old who present with an acute febrile illness that is clinically suggestive of bacteremia.
Sampling Method: Non-Probability Sample
Enrollment: 969 (Actual)
Dates: Start 2012-09-13 (Actual); Primary Completion 2017-03-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Typhoid fever-specific host response classifier genes | 10 years
  Define typhoid fever-specific host response classifier genes using gene expression (GE) micro-arrays.
Serum anti-typhoid fever proteins | 10 years
  Discover specific serum anti-typhoid fever proteins using newly established S. Typhi proteome micro-arrays and develop prototype serologic assay for acute typhoid (ELISA)
Validate classifier genes and field-test prototype ELISAs | 10 years
  Validate classifier genes and field-test prototype ELISAs using new, independent cohorts.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen K Obaro, MD, Principal Investigator — Univeristy of Nebraska Medical Center
Locations (1):
- National Hospital of Nigeria, Abuja, Nigeria